CLINICAL TRIAL: NCT00406198
Title: Phase 4 Randomized Multicentric Controlled Study on Impact of Continuous Venovenous Hemofiltration on Organ Failure at the Early Phase of Severe Sepsis
Brief Title: Impact of Continuous Venovenous Haemofiltration on Organ Failure During the Early Phase of Severe Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Collaborators: Ministry of Health, France (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DP 97 02 06; ministère recherche EA 322
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Bacteremia; Gram-Negative Bacterial Infections; Gram-Positive Bacterial Infections; Pneumonia, Bacterial; Shock, Septic; Sepsis
Keywords: Sepsis syndrom; severe sepsis; septic shock; hemofiltration; multiple organ failure
MeSH Terms: conditions — Bacteremia; Gram-Negative Bacterial Infections; Gram-Positive Bacterial Infections; Pneumonia, Bacterial; Shock, Septic; Sepsis; Multiple Organ Failure | interventions — Hemofiltration

INTERVENTIONS:
Procedure: venovenous hemofiltration

SUMMARY:
The impact of continuous veno-venous haemofiltration (CVVH) on sepsis-induced multiple organ failure severity is controversial. We thus sought to assess the effect of early application of haemofiltration on the degree of organ dysfunction and plasma cytokine levels in patients with severe sepsis or septic shock.

DETAILED DESCRIPTION:
prospective, randomized, open, multicentre study was performed between 1997 and 1999 in 16 French intensive care units. Patients were enrolled within 24 hours of development of the first organ failure related to a new septic insult. They were randomized to group 1 (HF), who received haemofiltration for a 96 hr period, or group 2 (C) who were managed conventionally. The primary end-point was the number, severity and duration of organ failures at 14 days, as evaluated by the SOFA score, on an intention-to-treat analysis. Strict guidelines were provided to perform continuous haemofiltration under the same conditions and objectives in all centres.

ELIGIBILITY:
Inclusion Criteria:

* clinically identified focus of infection associated with at least 2 SIRS criteria and one or more sepsis-induced organ failures within the 24 hours prior to inclusion, plus a SAPS II score between 35-63

Exclusion Criteria:

* Patients were excluded if pregnant, younger than 18 years, in a moribund state, in chronic renal failure, or receiving immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1997-03; Study Completion 1999-12

PRIMARY OUTCOMES:
The primary end-point was the number, severity and duration of organ failures at 14 days, as evaluated by the SOFA score, on an intention-to-treat analysis

SECONDARY OUTCOMES:
Secondary end point : safety, ventilation and hemodynamic support weaning

CONTACTS AND LOCATIONS:
Overall Officials: Didier Payen, MD, PhD, Principal Investigator — Hpopital Lariboisiere
Locations (1):
- Lariboisiere University Hospital, Paris, France